CLINICAL TRIAL: NCT01060150
Title: Efficacy and Learning Skill After OROS Methylphenidate Treatment in Adolescents With Attention-Deficit/Hyperactivity Disorder: A 12-week, Multi-center, Open-label Study
Brief Title: An Efficacy Study of Osmotic Release Oral System (OROS) Methylphenidate in Participants With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015496; CON-KOR-4019; CONCERTAATT4082
Record Dates: First submitted 2010-01-21; First posted 2010-02-02 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate hydrochloride; Methylphenidate; CONCERTA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OROS Methylphenidate HCl (Experimental)
  Interventions: Drug: OROS Methylphenidate HCl

INTERVENTIONS:
Drug: OROS Methylphenidate HCl — Osmotic Release Oral System (OROS) Methylphenidate HCl tablet will be given orally once daily at a starting dose of 18 milligram (mg) for those less than 30 kilogram (kg) of body weight and 27 mg for those more than or equal to 30 kg; the dose can be increased by 9 mg or 18 mg per week up to Week 6 depending on a participant's treatment effect and tolerability; then a maximum maintenance dose of 72 mg will be given orally once daily up to Week 12.
  Other Names: Concerta

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and effects of Osmotic Release Oral System (OROS) methylphenidate hydrochloride (HCl) on learning skill changes in Korean participants with Attention-Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This is 12 week, open label (all people involved know the identity of the intervention), prospective (study following participants forward in time), single arm, multicenter study (when more than one hospital or medical school team work on a medical research study) of OROS methylphenidate HCl. The study will consist of 6 visits at Screening, Baseline, Week 1, 3, 6 and 12. The participants already on other ADHD medications in addition to methylphenidate will be required to undergo a washout period (period when receiving no treatment) of at least 1 week. The participants will be on once daily study medication starting at 18 milligram per day (mg/day) in participants with less than 30 kilogram (kg) of body weight or at 27 mg/day in participants with more than 30 kg. The dose will be increased by 9 mg or 18 mg every week for up to Week 6 based on the treatment efficacy and tolerability, followed by a maximum maintenance dose of 72 mg orally once daily up to Week 12, during which the dose can be decreased by 9 mg depending on tolerability. Efficacy will primarily be assessed using Clinical Global Impression of Severity of Illness (CGI-S) scale, Clinical Global Impression of Improvement of Illness (CGI-I) scale, Korean version of ADHD-IV Rating Scale (K-ARS) and Learning Skill Test (LST) score. Participants' safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for Attention Deficit Hyperactivity Disorder (ADHD) and are considered to require medication therapy
* Participants that agreed to observe visit schedules and willingly complete the evaluation defined by participant (possibly to be completed by parents/guardians) during the treatment period
* Participants and parents/guardians that are able to understand the participation procedures of the research and spontaneously request the discontinuation therein at any time
* Participants that offered spontaneous consent for participation
* Participants whose guardian/legal representative provided spontaneous written consent

Exclusion Criteria:

* Hypersensitivity to methylphenidate HCl
* Participants diagnosed with major depression or anxiety disorders according to DSM-IV Diagnostic criteria and who requires drug therapy
* Participants with a history of bipolar disorder, psychotic disorder, and substance abuse disorder ordiagnosed with an overall developmental disorder, organic brain disorder, seizure (sudden, uncontrolled muscle spasms and loss of consciousness resulting from abnormal brain function) disorder, movement disorder requiring the medication therapy, or with a family history of Tourette's syndrome (a neuropsychological disorder that causes marked distress or significant impairment in social, occupational, or other important areas of functioning)
* Taken Osmotic Release Oral System (OROS) Methylphenidate within 3 months prior to screening
* Currently taking alpha-2 adrenergic receptor agonist, antidepressant, antipsychotic, benzodiazepines, modafinil, anticonvulsant (drug used to stop seizures) or health food supplements that may have a central nervous system activity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- [Derived] Na KS, Lee SI, Hong SD, Kim JH, Shim SH, Choi J, Yang J, Lee MS, Joung YS, Kim EJ, Park JH. Effect of osmotic-release oral system methylphenidate on learning skills in adolescents with attention-deficit/hyperactivity disorder: an open-label study. Int Clin Psychopharmacol. 2013 Jul;28(4):184-92. doi: 10.1097/YIC.0b013e3283612509. PMID 23587983

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS Methylphenidate HCl: Osmotic Release Oral System (OROS) Methylphenidate hydrochloride (HCl) tablet orally once daily at a starting dose of 18 milligram (mg) for those less than 30 kilogram (kg) and 27 mg for those more than or equal to 30 kg; the dose could be increased by 9 mg or 18 mg per week up to Week 6 depending on a participant's treatment effect and tolerability; then a maximum maintenance dose of 72 mg orally once daily up to Week 12
Period: Overall Study
Arm/Group | OROS Methylphenidate HCl
Started | 115
Treated | 113
Completed | 92
Not Completed | 23
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 8
Not completed — Enrolled, but not treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 113
Age Continuous [Mean (Standard Deviation); unit: Years] | 15.24 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 86
Korean Version of Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (K-ARS) Score [Mean (Standard Deviation); unit: Units on a scale] — The K-ARS is a rating scale that is used for the ADHD diagnosis and the assessment of treatment efficacy and comprises 18 items in total on the basis of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), each item being rated from 0-3 points. The total score ranges from 0-54 with higher score indicating more severity of the condition.
  Units on a scale | 27.58 (8.92)
Clinical Global Impression - Severity (CGI-S) Score [Mean (Standard Deviation); unit: Units on a scale] — The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
  Units on a scale | 4.88 (0.79)
Learning Skill Test (LST) Total Score [Mean (Standard Deviation); unit: T-score] — The LST measures learning ability of student. It is composed of 7 sections: self control, participation, task accomplishment, reading, writing, test taking and information processing. It consists of 70 items for middle school student and 80 items for high school student. Each item is rated on 5-point Likert scale (1=never to 5=always). Total score range:70-350 (middle school) and 80-400 (high school). In result analysis, each sub-score and total score was converted to T-score for normalization. Score range of T-score: 1-100 with a mean of 50. Higher score indicates better ability for learning.
  T-score | 40.97 (11.07)

OUTCOME MEASURES:

1. Primary Outcome: Korean Version of the Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (K-ARS) Score
Description: The K-ARS is a rating scale that is used for the ADHD diagnosis and the assessment of treatment efficacy and comprises 18 items in total on the basis of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), each item being rated from 0-3 points. The total score ranges from 0-54 with 0=normal and 54=severe condition.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants who received the study drug at least once, satisfied the inclusion and exclusion criteria, and had efficacy assessment data at the Baseline. Missing values at Week 12 were imputed using Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 113
Units on a scale | 11.78 (7.64)

2. Primary Outcome: Clinical Global Impression - Severity (CGI-S) Score
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Week 12
Population: ITT population included all participants who received the study drug at least once, satisfied the inclusion and exclusion criteria, and had efficacy assessment data at the Baseline. Missing values at Week 12 were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 113
Units on a scale | 2.81 (1.12)

3. Primary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 12
Population: ITT population included all participants who received the study drug at least once, satisfied the inclusion and exclusion criteria, and had efficacy assessment data at the Baseline. Here 'N' (Number of Participants Analyzed) represents number of participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 103
Units on a scale | 2.14 (0.75)

4. Primary Outcome: Learning Skill Test (LST) Total Score
Description: The LST measures learning ability of student. This scale is composed of 7 sections: self control, participation, task accomplishment, reading, writing, test taking and information processing. It consists of 70 items for middle school student (age 13-15 years) and 80 items for high school student (age 16-18 years). Each item is rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The total score range is 70-350 for middle school version and 80-400 for high school version where higher score indicates better ability for learning. In result analysis, each sub-score and total score was converted to T-score for normalization. The score range of T-score is from 1 to 100 with a mean of 50. Higher score indicates better ability for learning.
Time Frame: Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 98
T-score | 49.61 (11.57)

5. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder (ADHD) Diagnostic System (ADS) Test Result for Omission Errors and Commission Errors
Description: The ADS is composed of 4 factors: omission/missing frequency to measure attention dispersibility; false alarm/commission frequency to measure impulse; mean response/reaction time to measure the speed of task processing; and the response variability/standard deviation of response time to measure the consistency of attention. The total value for both, omission errors and commission errors, ranges from 0-100 errors where high value indicates worsening attention.
Time Frame: Baseline and Week 12
Population: The ITT population included all participants who received the study drug at least once, satisfied the inclusion and exclusion criteria, and had efficacy assessment data at the Baseline. Here 'N' (Number of Participants Analyzed) represents number of participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 101
Errors
  Omission errors: Baseline | 58.88 (27.35)
  Omission errors: Week 12 | 57.40 (48.79)
  Commission errors: Baseline | 62.98 (32.32)
  Commission errors: Week 12 | 51.70 (21.19)

6. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder (ADHD) Diagnostic System (ADS) Test Score for Reaction Time and Response Variability
Description: The ADS is composed of 4 factors: omission/missing frequency to measure attention dispersibility; false alarm/comission frequency to measure impulse; mean response/reaction time to measure the speed of task processing; and the response variability/standard deviation of response time to measure the consistency of attention. The score range for both, reaction time and response variability, is 0-100. High score indicates worsening attention. If one or over factor's score is over 65 point, the participant is resulted in having attention deficit.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 101
Units on scale
  Reaction time average: Baseline | 54.32 (15.45)
  Reaction time average: Week 12 | 49.73 (26.33)
  Response variability: Baseline | 85.77 (60.21)
  Response variability: Week 12 | 59.42 (64.77)

7. Secondary Outcome: Digit Span Test Score
Description: Each participant individually was given a sequence of numbers, with the sequence becoming progressively longer, to repeat the digits in the same sequence, either forwards or backwards. Each sequence length was attempted twice. The test was complete after failure on both trials of any sequence length. 1 point was awarded if the participant passed only 1 trial of a sequence length. 0 points were given if the participant failed both trials. Total score range was 0-16 (forwards) and 0-14 (backwards). A higher score was indicative of better recall and attention.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Units on a scale
  Forward: Baseline | 11.19 (2.92)
  Forward: Week 12 | 11.56 (2.90)
  Backward: Baseline | 7.09 (2.39)
  Backward: Week 12 | 7.32 (2.41)

8. Secondary Outcome: Finger Window (FW) Test Score
Description: In FW test, a participant shows memory of a demonstrated visual pattern using a 8x11 inch plastic template containing 9 asymmetrically located holes. The examiner models a given sequence of holes and asks the participant to imitate the sequence by placing his/her finger through the same holes in the correct order. The total number of correct sequences constitutes the total score which ranges from 0-24 (forward FW) and 0-28 (backward FW) with higher score indicating a more favorable health state.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Units on a scale
  Forward FW: Baseline | 18.42 (4.60)
  Forward FW: Week 12 | 19.09 (4.49)
  Backward FW: Baseline | 15.59 (4.97)
  Backward FW: Week 12 | 17.36 (3.84)

9. Secondary Outcome: Controlled Oral Words Association Test (COWAT) Score
Description: This test measures the executive function of the frontal lobe and is consisted of examinations of category/meaning fluency and letter/phoneme fluency. It consisted of three 60 second word generation trials in which the participant orally generates as many words as possible that begin with target letters F, A and S. Dependent variables included total number of acceptable words generated for each target letter and total number of words generated across all three letter trials. Total score was calculated as sum of acceptable words generated, with higher scores indicating better verbal fluency.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Words
  Category/semantic: Baseline | 29.71 (5.86)
  Category/semantic: Week 12 | 30.62 (6.16)
  Letter/phenomic: Baseline | 28.71 (10.82)
  Letter/phenomic: Week 12 | 33.78 (11.18)

10. Secondary Outcome: Stroop Test Result for Reaction Time
Description: This test consists of 3 trials: color trial (simple execution), word trial (middle execution) and word-color interference trial (interfering execution). In simple execution, participants have to read the written color names of the words independent of the color of the ink. In middle execution, participants have to read words written in black letters. In interfering experiment, participants have to say the color of the letters independent of the written word. This test estimates spending time for execution. High spending time indicates low ability of suppression of automation.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Seconds
  Simple execution time: Baseline | 14.78 (3.8)
  Simple execution time: Week 12 | 13.64 (3.27)
  Middle execution time: Baseline | 15.88 (3.56)
  Middle execution time: Week 12 | 15.04 (4.57)
  Interfering execution time: Baseline | 22.12 (6.18)
  Interfering execution time: Week 12 | 19.72 (5.63)

11. Secondary Outcome: Stroop Test Result for False Reaction
Description: This test consists of 3 trials: color trial (simple execution), word trial (middle execution) and word-color interference trial (interfering execution). In simple execution, participants have to read the written color names of the words independent of the color of the ink. In middle execution, participants have to read words written in black letters. In interfering experiment, participants have to say the color of the letters independent of the written word. The total value ranges from 0-24 errors for each execution where high value indicates worsening attention.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Errors
  Simple execution false reaction: Baseline | 0.4 (0.77)
  Simple execution false reaction: Week 12 | 0.16 (0.39)
  Middle execution false reaction: Baseline | 0.3 (0.67)
  Middle execution false reaction: Week 12 | 0.2 (0.47)
  Interfering execution false reaction: Baseline | 1.04 (1.29)
  Interfering execution false reaction: Week 12 | 0.84 (1.00)

12. Secondary Outcome: Stroop Test Score for Ratio Interference
Description: Ratio interference is calculated by dividing simple execution time by interfering execution time. The score range is 0-1. Higher value indicates better ability of suppression of automation.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Methylphenidate HCl
Number analyzed (Participants) | 100
Units on a scale
  Baseline | 0.70 (0.19)
  Week 12 | 0.72 (0.19)

ADVERSE EVENTS:
Time Frame: After signing of informed consent up to Week 12
Arm/Group | OROS Methylphenidate HCl
Serious Adverse Events (participants affected / at risk) | 2/113
Other Adverse Events (participants affected / at risk) | 98/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Methylphenidate HCl (N=113)
Lymphadenitis (Blood and lymphatic system disorders) | 1
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Methylphenidate HCl (N=113)
Decreased appetite (Metabolism and nutrition disorders) | 66
Nausea (Gastrointestinal disorders) | 32
Abdominal pain upper (Gastrointestinal disorders) | 19
Stomach discomfort (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Insomnia (Psychiatric disorders) | 37
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 9
Nervousness (Psychiatric disorders) | 7
Anger (Psychiatric disorders) | 6
Headache (Nervous system disorders) | 31
Dizziness (Nervous system disorders) | 11
Somnolence (Nervous system disorders) | 8
Irritability (General disorders) | 16
Fatigue (General disorders) | 13
Nasopharyngitis (Infections and infestations) | 19
Palpitations (Cardiac disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less